CLINICAL TRIAL: NCT03509961
Title: A Phase II Pilot Trial to Estimate Survival After a Non-total Body Irradiation (TBI) Based Conditioning Regimen in Patients Diagnosed With B-acute Lymphoblastic Leukemia (ALL) Who Are Pre-allogeneic Hematopoietic Cell Transplantation (HCT) Next-generation-sequence (NGS) Minimal Residual Disease (MRD) Negative
Brief Title: The EndRAD Trial: Eliminating Total Body Irradiation (TBI) for NGS-MRD Negative Children, Adolescents, and Young Adults With B-ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pediatric Transplantation & Cellular Therapy Consortium (Other)
Responsible Party: Principal Investigator, Michael Pulsipher, Principal Investigator, Children's Hospital Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-18-00141
Record Dates: First submitted 2018-03-19; First posted 2018-04-27 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2024-11

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Observational Arm (Other): Patients are enrolled to the observational arm to proceed with NGS-MRD testing pre-HCT. If NGS-MRD negative, eligible patients may be considered for the Treatment Arm to receive a myeloablative non-TBI conditioning regimen prior to HCT.
  If NGS-MRD positive, patients may continue in the observational arm and receive HCT under the direction of their transplant physician and followed on the study for outcome.
  Interventions: Diagnostic Test: NGS-MRD
- Treatment Arm (Other): Patients enrolled to the observational arm that are NGS-MRD pre-HCT are considered for the Treatment Arm. Patients will receive a myeloablative non-TBI conditioning regimen prior to the transplant consisting on busulfan, fludarabine and thiotepa. Patients will be followed for outcome for up to 5 years.
  Interventions: Diagnostic Test: NGS-MRD; Drug: Myeloablative allogeneic HCT with a non-TBI conditioning regimen

INTERVENTIONS:
Diagnostic Test: NGS-MRD — Next generation sequencing minimal residual disease (NGS-MRD) is a test that has increased sensitivity over multichannel flow cytometry to better identify risk of key outcomes after HCT. Patients that have a pre-HCT negative NGS-MRD results may be eligible to proceed to the treatment arm of the study that uses a non-TBI conditioning regimen.
Drug: Myeloablative allogeneic HCT with a non-TBI conditioning regimen — Myeloablative study regimen will consist of busulfan, fludarabine and thiotepa.
  day -7: Fludarabine and Busulfan day -6: Fludarabine and Busulfan day -5: Fludarabine and Busulfan day -4: Fludarabine and Busulfan day -3: Fludarabine day -2: Thiotepa day -1: Rest Day 0: Transplant
  Arms: Treatment Arm

SUMMARY:
This study will evaluate the use of non- TBI (total body irradiation) conditioning for B-ALL patients with low risk of relapse as defined by absence of NGS-MRD (next generation sequencing minimal residual disease) before receiving a hematopoietic cell transplant (HCT). Patients diagnosed with B-ALL who are candidates for HCT will be screened by NGS-MRD on a test of bone marrow done before the HCT. Subjects who are pre-HCT NGS-MRD negative will be eligible to receive a non-TBI conditioning regimen as part of the treatment cohort of the study. Subjects who are pre-HCT NGS-MRD positive will be treated as per treating center standard and will be followed in an observational cohort (HCT center standard of care).

DETAILED DESCRIPTION:
A Phase II pilot trial will estimate survival after a non-TBI based conditioning regimen in patients diagnosed with B-acute lymphoblastic leukemia (ALL) who are pre-allogeneic hematopoietic cell transplantation (HCT) next-generation-sequence (NGS) minimal residual disease (MRD) negative.

The relationship of NGS-MRD status to survival in children, adolescents, and young adults with B-ALL undergoing any approach to allogeneic HCT will be explored in a larger cohort (treatment [phase II] and observational arms of the study).

The primary objective is to estimate 2-year event free survival (EFS) in pre-HCT NGS-MRD negative patients with B-ALL undergoing a non-TBI based conditioning regimen through a multi-center prospective trial. The accrual period is 3 years.

Patients that are NGS-MRD negative with B-ALL may be eligible for the Treatment Arm, which is myeloablative non-TBI conditioning with busulfan, fludarabine, and thiotepa followed -matched related, unrelated, and umbilical cord blood transplants. Patients that are NGS-MRD positive will be followed on the observational arm for outcome.

Study sampling will include NGS-MRD bone marrow (BM) aspirate and peripheral blood (PB) samples collected [same day when possible] pre-HCT (within 4 weeks), and post-HCT on days 42 ± 14, 100 ± 20, and 365 ± 60; PB samples only will also be collected day 180± 60 and 270± 60; day +30, day +100, and 1-year post-HCT. NGS-MRD peripheral blood sample only at 6 months and 9 months post-HCT; (Blast specimen at time of diagnosis or relapse is required for NGS-MRD testing).

ELIGIBILITY:
Inclusion Criteria for the Observational Arm:

Any patient with ALL who undergoes Myeloablative HCT including any of the following:

* Patients who are pre-HCT NGS-MRD positive.
* Patients <1 year old who are pre-HCT NGS-MRD negative.
* Patients who are pre-HCT NGS-MRD negative (CR1/CR2) who received inotuzumab ozogamicin therapy before proceeding to HCT.
* Patients who are pre-HCT NGS-MRD negative and will be receiving haploidentical HCT.
* Patients who are pre-HCT NGS-MRD negative in CR2 with history of CNS relapse.
* Patients who have received blinatumomab, but are >CR2 prior to HCT.
* Patients who have received CART-T cellular therapy, but are >CR2 prior to HCT.
* Patients with pre-HCT NGS-MRD negative in ≥ CR3.
* Any T-ALL and MPAL patients undergoing first allogeneic HCT
* Any patient who is pre-HCT NGS-MRD negative and eligible for participation in the treatment arm but family does not consent for treatment arm or treating physician believe it is in the patient best interest not to enroll on the treatment arm

Inclusion Criteria for the Treatment Arm:

* Pre-HCT NGS-MRD negative
* Age ≥ 1 year and ≤ 25 years
* Disease status: B-ALL in first (CR1) or second remission (CR2)
* No prior allogeneic hematopoietic stem cell transplant.
* Patients in CR1 or CR2 after blinatumomab treatment.
* Patients in CR1 or CR2 after CAR-T cellular therapy.
* Karnofsky Index or Lansky Play-Performance Scale ≥ 60 % on pre-transplant evaluation. Karnofsky scores must be used for patients > 16 years of age and Lansky scores for patients < 16 years of age.
* Able to give informed consent if > 18 years, or with a legal guardian capable of giving informed consent if < 18 years.
* Adequate organ function (within 4 weeks of initiation of preparative regimen), defined as:
* Pulmonary: FEV1, FVC, and corrected DLCO must all be ≥ 50% of predicted by pulmonary function tests (PFTs). For children who are unable to perform for PFTs due to age, the criteria are: no evidence of dyspnea at rest and no need for supplemental oxygen.
* Renal: Creatinine clearance or radioisotope GFR ≥ 60 mL/min/1.73 m2 or a serum creatinine based on age/gender.
* Cardiac: Shortening fraction of ≥ 27% by echocardiogram or radionuclide scan (MUGA) or ejection fraction of ≥ 50% by echocardiogram or radionuclide scan (MUGA), choice of test according to local standard of care.
* Hepatic: SGOT (AST) or SGPT (ALT) < 5 x upper limit of normal (ULN) for age. Conjugated bilirubin < 2.5 mg/dL, unless attributable to Gilbert's Syndrome.

Exclusion Criteria:

* CR2: exclude patients with history of CNS relapse (i.e. in CR2 with history of CNS isolated or combined relapse; CNS 2 will also be considered as CNS 3 for this purpose) from the treatment arm of study (can be enrolled on the observational arm).
* Patients who have received inotuzumab treatment prior to allogeneic HCT are NOT eligible for the study treatment arm. Inotuzumab treatment may increase the risk of VOD/SOS for any allogeneic HCT recipient, but could potentiate the risk for with busulfan-based myeloablation (study-directed non-TBI conditioning). All inotuzumab-treated patients are eligible for the observational arm (HCT center standard of care).
* Patients receiving non-myeloablative conditioning are not allowed on the observational arm (reduced toxicity conditioning with Flu/Mel/Thio is allowed on the observational arm).
* Pregnant or lactating females are ineligible as many of the medications used in this protocol could be harmful to unborn children and infants.
* Patients with HIV or uncontrolled fungal, bacterial or viral infections are excluded. Patients with history of fungal disease during induction therapy may proceed if they have a significant response to antifungal therapy with no evidence or minimal evidence of non-progressive disease remaining by CT evaluation.
* Patients with active CNS leukemia or any other active site of extramedullary disease at the time of enrollment are not permitted.
* T-ALL and MPAL patients are only allowed on the observational arm.
* Patients with genetic disorders (generally marrow failure syndromes) prone to secondary AML/ALL with known poor outcome are not eligible (Fanconi Anemia, Kostmann Syndrome, Dyskeratosis Congenita, etc).

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Estimated)
Dates: Start 2018-08-29 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Two Year Event-free Survival | Two years
  The primary objective of this study is the two Year Event-free Survival for patients with high-risk or recurrent B-ALL who proceed to HCT and who are NGS-MRD negative when treated with a non-TBI preparative regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Abdel-Azim Hisham, MD, Principal Investigator — Loma Linda University; Troy Quigg, DO, MS, Principal Investigator — Helen DeVos Children's Hospital
Locations (24):
- United States (24):
  - Children's of Alabama/University of Alabama in Birmingham(UAB), Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - City of Hope, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCLA Mattel Children's Hospital, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - UCSF, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Alfred I. duPont Hospital for Children - Nemours Deleware, Wilmington, Delaware
  - University of Florida, Gainesville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Riley Hospital for Children - Indiana University, Indianapolis, Indiana
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - Dana Faber Cancer Institute/ Boston Children's Hospital, Boston, Massachusetts
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Children's Mercy Hospital, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Atrium Health - Levine Cancer Center, Charlotte, North Carolina
  - The University of Texas M. D. Anderson Cancer Center, Houston, Texas
  - Methodist Healthcare System, San Antonio, Texas

REFERENCES:
- [Derived] Andolina JR, Fries C, Boulware R, Vargas A, Fraint E, Barth M, Ambrusko S, Comito M, Monteleone P. Successful Bone Marrow Transplantation With Intensive Post-transplant Intrathecal Chemotherapy for CNS Relapsed AML in 2 Infants. J Pediatr Hematol Oncol. 2022 Jan 1;44(1):e264-e267. doi: 10.1097/MPH.0000000000002151. PMID 33843815